CLINICAL TRIAL: NCT00075907
Title: A Comparative Trial of Protease-Containing and Protease-Sparing HAART Regimens in HIV-Infected Adolescents With an Evaluation of Therapeutic Drug Monitoring
Brief Title: Anti-HIV Drug Regimens With or Without Protease Inhibitors and Drug Level Monitoring in HIV Infected Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACTG P1034; DAIDS-ES ID 10043
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Lopinavir; Ritonavir

INTERVENTIONS:
Drug: Efavirenz + 2 NRTIs
Drug: Lopinavir/Ritonavir + 2 NRTIs
Procedure: Therapeutic Drug Monitoring

SUMMARY:
The purpose of this study is to compare the effectiveness of anti-HIV drug regimens with or without a protease inhibitor (PI) in HIV infected adolescents. It will also determine if monitoring drug levels and adjusting the dose as necessary improves the effectiveness of these regimens.

DETAILED DESCRIPTION:
HIV infected adolescents may have a significantly higher capacity for immune reconstitution following highly active antiretroviral therapy (HAART), compared to adults. Despite this advantage, HIV infected adolescents are often reluctant to get proper medical care, follow through with doctor appointments, and adhere to medication schedules and regimens necessary to keep their infection under control. Lopinavir/ritonavir (LPV/r), a PI, and efavirenz (EFV), a non-nucleoside reverse transcriptase inhibitor (NNRTI), both have long half-lives that make them ideal drugs for the adolescent population, as they are more forgiving if patients miss or sleep through doses. The availability of once-daily dosing of LPV/r will reduce pill burden and offers more flexibility in medication scheduling, also helping to promote treatment adherence among this age group. This study will examine the effectiveness of two HAART regimens, one with the PI LPV/r and two nucleoside reverse transcriptase inhibitors (NRTIs), and the other with the NNRTI EFV and two NRTIs. The efficacy of therapeutic drug monitoring (TDM) and subsequent dose adjustment will also be assessed with both regimens.

Patients will be enrolled in this study for 96 weeks and will be randomly assigned into one of two groups. Group 1 will receive LPV/r and 2 NRTIs. Treatment naive patients in Group 1 will have the option of receiving either once-daily dosing or twice-daily dosing of LPV/r. Treatment experienced patients will receive twice-daily dosing of LPV/r. Patients on once-daily dosing of LPV/r who become intolerant to the regimen will be permitted to switch to twice-daily dosing. Group 2 will receive EFV and 2 NRTIs. All patients will be independently and simultaneously randomly assigned to undergo either TDM with subsequent dose adjustment if necessary or no TDM.

Patient medical history and physical exam will be conducted at screening, entry, Weeks 2, 4, 8, every 8 weeks until Week 48, and every 12 weeks thereafter. Blood collection will occur at all study visits. Self-reported pill counts and MEMS TrackCap readings (on LPV/r and EFV bottles) will be noted at most visits. Patients will be asked to complete adherence questionnaires at selected study visits.

Patients enrolled in PACTG 390 (Different Combination Regimens and Treatment-Switching Guidelines in HIV Infected Children 18 Years of Age and Younger) are encouraged to coenroll simultaneously in this study and in PACTG 219C (Long-Term Effects of HIV Exposure and Infection in Children).

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* HIV RNA viral load of 10,000 copies/ml or more at screening
* Weigh 35 kg (77.2 lbs) or more
* HAART naive or received a single regimen of combination therapy consisting of NRTIs with or without a single PI (except LPV). Patients who received zidovudine monotherapy during pregnancy or used low-dose ritonavir (RTV) as a PI boost are not excluded.
* For PI experienced patients, have sensitivity to LPV at screening
* Able to receive, as part of background HAART chosen by their physician, at least one new NRTI that is likely to be active against the patient's virus and unlikely to have cross-resistance with previously used NRTIs
* Willing to use acceptable forms of contraception
* Parent or legal guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Prior receipt of any NNRTI or LPV
* Require certain medications
* Grade 3 or 4 clinical or laboratory toxicity, as defined by the Division of AIDS Toxicity Table for Grading Severity of Pediatric Adverse Effects
* Chemotherapy for active malignancy
* Acute opportunistic or serious bacterial infection requiring therapy at study entry
* Investigational treatment within 30 days of study entry
* Score of 20 or more on Beck Depression Inventory (BDI-II) or suicidal thoughts on BDI-II (score of 2 or 3 on Question 9), regardless of total score
* Pregnant within 48 hours of starting EFV
* Breastfeeding

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240
Dates: Start 2004-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving viral suppression (viral load less than 1,000 copies/ml) at Week 24 and maintaining suppression through Week 48 while remaining on study treatment

SECONDARY OUTCOMES:
Proportion of patients achieving virologic suppression (viral load less than 1,000 copies/ml) at Week 24 and maintaining suppression through Week 96 while remaining on study treatment
adherence measured by MEMS TrackCap Monitors (percentage of doses taken, estimated using the frequency of bottle openings recorded by the MEMS TrackCap Monitors, the MEMS TrackCap Monitor tracking form, and the information recorded on the questionnaires)
adherence measured by patient self-report (binary variable of perfect adherence measured 3 days prior to any study visit reported on the adherence questionnaires and the numbers of visits with reported perfect adherence up to Week 24, 48, and 96)
adherence measured by pill count (percentage of pills taken, determined by counting the pills left in the bottles)
HIV viral load at each study visit
number and severity of symptoms of distress and central nervous system (CNS) side effects
number and severity of all adverse events of Grade 3 or more attributed to study treatment
time to virologic failure (first time viral load is measured to be 1,000 copies/ml or more after Week 24, time before discontinuing study treatment for any reason before Week 96, or time before terminating study for any reason before Week 96)
HIV resistance mutations at baseline and at time of virologic failure (viral load returning to 1,000 copies/ml or more)
baseline values for percentage and total number of CD19 (B cells), total T cells (CD3 T cells), CD4 (T helper cells), CD8 (cytotoxic T cells), naive CD4 T cells (CD62L/CD45RA/CD4), and activated CD8 T cells (HLADR/CD38/CD8)
changes from baseline to Weeks 24, 48, and 96 for percentage and total number of CD19 (B cells), total T cells (CD3 T cells), CD4 (T helper cells), CD8 (cytotoxic T cells), naive CD4 T cells (CD62L/CD45RA/CD4), and activated CD8 T cells (HLADR/CD38/CD8)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Silio, MD, Study Chair — Tulane Medical Center; Russell Van Dyke, MD, Study Chair — Tulane Medical Center
Locations (13):
- United States (13):
  - Usc La Nichd Crs, Alhambra, California
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Children's Hospital of Los Angeles NICHD CRS, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Children's Hosp., New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Children's Med. Ctr. Dallas, Dallas, Texas
  - Texas Children's Hosp. CRS, Houston, Texas

REFERENCES:
- [Background] Eron JJ, Feinberg J, Kessler HA, Horowitz HW, Witt MD, Carpio FF, Wheeler DA, Ruane P, Mildvan D, Yangco BG, Bertz R, Bernstein B, King MS, Sun E. Once-daily versus twice-daily lopinavir/ritonavir in antiretroviral-naive HIV-positive patients: a 48-week randomized clinical trial. J Infect Dis. 2004 Jan 15;189(2):265-72. doi: 10.1086/380799. Epub 2004 Jan 7. PMID 14722892
- [Background] Deschamps AE, Graeve VD, van Wijngaerden E, De Saar V, Vandamme AM, van Vaerenbergh K, Ceunen H, Bobbaers H, Peetermans WE, de Vleeschouwer PJ, de Geest S. Prevalence and correlates of nonadherence to antiretroviral therapy in a population of HIV patients using Medication Event Monitoring System. AIDS Patient Care STDS. 2004 Nov;18(11):644-57. doi: 10.1089/apc.2004.18.644. PMID 15633262
- [Background] Murphy DA, Sarr M, Durako SJ, Moscicki AB, Wilson CM, Muenz LR; Adolescent Medicine HIV/AIDS Research Network. Barriers to HAART adherence among human immunodeficiency virus-infected adolescents. Arch Pediatr Adolesc Med. 2003 Mar;157(3):249-55. doi: 10.1001/archpedi.157.3.249. PMID 12622674
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Van Dyke RB, Lee S, Johnson GM, Wiznia A, Mohan K, Stanley K, Morse EV, Krogstad PA, Nachman S; Pediatric AIDS Clinical Trials Group Adherence Subcommittee Pediatric AIDS Clinical Trials Group 377 Study Team. Reported adherence as a determinant of response to highly active antiretroviral therapy in children who have human immunodeficiency virus infection. Pediatrics. 2002 Apr;109(4):e61. doi: 10.1542/peds.109.4.e61. PMID 11927734
- See also: Click here for more information about PACTG 390 — http://clinicaltrials.gov/ct/show/NCT00039741
- See also: Click here for more information about PACTG 219C — http://clinicaltrials.gov/ct/show/NCT00006304